CLINICAL TRIAL: NCT06076187
Title: Protein Digestion After Bariatric Surgery in Older Adults
Acronym: ProDigBO
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S67116
Record Dates: First submitted 2023-04-12; First posted 2023-10-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity; Bariatric Surgery Candidate; Aging; Protein Malabsorption
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group 1: Patients over 65 years of age who had undergone Roux-en-Y bariatric surgery: Group 1: Patients over 65 years of age who had undergone Roux-en-Y bariatric surgery
  Interventions: Other: Dual isotope protein digestibility method
- Group 2: Patients over 65 years of age who had undergone sleeve gastrectomy surgery: Group 2: Patients over 65 years of age who had undergone sleeve gastrectomy surgery
  Interventions: Other: Dual isotope protein digestibility method
- Group 3: Patients over 65 years of age without previous bariatric surgery: Group 3: Patients over 65 years of age without previous bariatric surgery
  Interventions: Other: Dual isotope protein digestibility method
- Group 4: Patients younger than 65 years of age who had undergone Roux-en-Y bariatric surgery: Group 4: Patients younger than 65 years of age who had undergone Roux-en-Y bariatric surgery
  Interventions: Other: Dual isotope protein digestibility method
- Group 5: Patients younger than 65 years of age who had undergone Sleeve Gastrectomy: Group 5: Patients younger than 65 years of age who had undergone Sleeve Gastrectomy
  Interventions: Other: Dual isotope protein digestibility method
- Group 6: Patients younger then 65 years of age without previous bariatric surgery: Group 6: Patients younger then 65 years of age without previous bariatric surgery
  Interventions: Other: Dual isotope protein digestibility method

INTERVENTIONS:
Other: Dual isotope protein digestibility method — Dual isotope method

SUMMARY:
The goal of this clinical trial is to investigate protein digestibility after bariatric surgery.

Does protein digestibility decrease after Roux-en-Y-Gastric Bypass? Does protein digestibility decrease after Sleeve Gastrectomy surgery? Does protein digestibility effect the ability to meet protein requirements?

DETAILED DESCRIPTION:
Purpose of clinical trial is to investigate the digestion of dietary protein in older patients who have undergone Roux-and-Y Bypass (RYGB) or sleeve gastrectomy (SG) surgery. The primary objective is to compare dietary protein digestion during a test meal who have previously undergone a RYGB surgery, SG surgery, or control patients, using a dual stable-isotope method. The secondary objectives are to investigate the relationship between protein intake corrected for protein digestion and skeletal muscle mass, and to investigate the relationship between the rate of free amino acid appearance and protein digestion.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Group 1,2,3: Age 65 years or older
* Group 4,5,6: Age 18 to 65 years
* Group 1,2,4,5: Previous bariatric surgery for obesity 1 - 10 years ago
* Group 3,6: No previous weight loss surgery

Exclusion Criteria:

* Current diagnosis of cancer
* Advanced organ failure, including chronic kidney disease Stage 5, liver cirrhosis Stage 3, intestinal failure, heart failure stage D, or chronic obstructive pulmonary disease stage 4.
* Immobility
* Neuromuscular degenerative conditions
* Gastrointestinal conditions including coeliac disease, Crohn's disease, previous resection of the small intestine, gastroparesis
* Unable to follow the procedures of the studies due to cognitive impairment such as diagnosed dementia.
* Allergy/intolerance to milk, or soy or spirulina

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with overweight, obesity or after bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
The proportion of dietary protein digested as measured by the dual-isotope method. | 3,5 hours
  The proportion of dietary protein digested as measured by the dual-isotope method.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Universitaire Ziekenhuizen KU Leuven, Leuven, Flemish Brabant
  - UZLeuven, Leuven, Vlaams Brabant

IPD SHARING:
Plan to Share IPD: Undecided